CLINICAL TRIAL: NCT03633006
Title: Blood Sample Collection in Subjects With Pulmonary Nodules or CT Suspicion of Lung Cancer or Pathologically Diagnosed Lung Cancer
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-01
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer (Diagnosis)
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood samples may be used for further analysis and future research. Samples may be stored for up to 20 years. These blood samples will be de-identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pulmonary Nodules: Subject with pulmonary nodules will be enrolled, provide a blood sample and may be followed up to 2 years for nodule resolution.
  A second blood draw will be collected at 12 months.
  Interventions: Other: Blood Sample Collection
- CT Suspicion of Cancer: Subject with suspicion of lung cancer will provide a blood sample.
  Diagnostic information will be collected to confirm the final diagnosis.
  Interventions: Other: Blood Sample Collection
- Pathologically Confirmed Cancer: Subject has pathologically confirmed lung cancer and is treatment naïve.
  Subject will be enrolled and provide a blood sample.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects participating in the study will have blood drawn at enrollment. Additional blood samples may be collected at 12 months from enrollment.
  Groups: Pulmonary Nodules
Other: Blood Sample Collection — Subjects participating in the study will have blood drawn at enrollment. Additional blood samples may be collected at 12 months from enrollment if lung cancer has not been confirmed.
  Groups: CT Suspicion of Cancer
Other: Blood Sample Collection — Subjects participating in the study will have blood drawn at enrollment.
  Groups: Pathologically Confirmed Cancer

SUMMARY:
The primary objective of this study is to obtain de-identified, clinically characterized, whole blood specimens for use in assessing new biomarkers for the detection of neoplasms of the lung. Subjects will be men and women, 35 years of age and older, with a CT confirmed nodule measuring 6-30 mm.

DETAILED DESCRIPTION:
Subjects with pulmonary nodules, a suspicion of lung cancer or pathologically confirmed, untreated lung cancer will be enrolled. Blood samples will be collected at enrollment and may be collected at 12 months for subjects with pulmonary nodules. Radiological and pathological data will be collected to confirm a cancer diagnosis or up to 2 years to assess nodule resolution.

ELIGIBILITY:
Inclusion Criteria:

* All Subjects:

  1. Subject is male or female, 35 years of age or older.
  2. Subject has at least one CT confirmed 6-30 mm nodule.
  3. Subject understands the study procedures and is able to provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

     Suspicion of Cancer Subjects:
  4. Subject has CT suspicion of lung cancer and is scheduled for biopsy or other diagnostic procedure.

Pathologically Confirmed Cancer Subjects:

4. Subject has pathologically confirmed lung cancer and is treatment naïve.

Pulmonary Nodule Subjects:

4. Subject has a recent (within 90 days of enrollment) CT radiological diagnosis of pulmonary nodule(s) without a scheduled biopsy/diagnostic procedure (other than CT or PET/CT).

Exclusion Criteria:

* All Subjects

  1. CT with IV contrast within 1 day [or 24 hours] of blood collection.
  2. Prior history of cancer within the past 5 years except for non-melanoma skin cancer. For subjects with suspicion of lung cancer who may have a concurrent work-up for another primary cancer, the non-lung cancer primary must be ruled out prior to enrollment.
  3. Prior removal of the lung, excluding percutaneous lung biopsy.
  4. Treatment (e.g., surgical resection, radiofrequency ablation) for pulmonary nodules prior to blood sample collection for this trial.
  5. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

     Pathologically Confirmed Cancer Subjects:
  6. Biopsy within 7 days prior to blood collection.
  7. Unresolved bleeding as a result of biopsy at the time of enrollment.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 3,250 subjects will be enrolled in this study. Subjects will be men and women, 35 years of age or older, with a CT confirmed nodule measuring 6-30 mm. Subjects will be enrolled into one of three groups: CT suspicion of lung cancer who are scheduled for biopsy/other diagnostic procedure; pathologically confirmed lung cancer that are treatment naïve; or recent positive CT showing pulmonary nodule(s) without a scheduled biopsy/diagnostic procedure.
Sampling Method: Non-Probability Sample
Enrollment: 3298 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Biomarker Identification | Subjects could be followed for up to 27 months.
  Screening subjects to find the appropriate methylation sites for the detection of lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Laura Strong, Study Director — Exact Sciences
Locations (83):
- United States (83):
  - Achieve Clinical Research, Birmingham, Alabama
  - Phoenix Medical Group, Peoria, Arizona
  - Newport NativeMD, Newport Beach, California
  - Palmtree Clinical Research, Inc, Palm Springs, California
  - Palo Alto Veterans Health Care, Palo Alto, California
  - Premier Medical Group, Upland, California
  - American Research Institute, Inc, Cutler Bay, Florida
  - International Research Partners, LLC, Doral, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Pulmonary Disease Specialists, Kissimmee, Florida
  - Medical Research of Central Florida, LLC, Leesburg, Florida
  - Future Clinical Research, Miami, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Orcinova AMS Research, Miami, Florida
  - Sunrise Research Institute, Inc, Miami, Florida
  - American Research Medical Group, Miami, Florida
  - Health and Life Research Institute, LLC, Miami, Florida
  - Care Research Center, Miami, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - AMPM research Clinic, Miami Gardens, Florida
  - Sarasota Memorial Hospital Clinical Research Center, Sarasota, Florida
  - Coastal Pulmonary and Critical Care, PLC, St. Petersburg, Florida
  - Pasadena Center for Medical Research, Inc, St. Petersburg, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Pulmonary Care Research Group, PA, Winter Park, Florida
  - Piedmont Healthcare, Inc., Atlanta, Georgia
  - Gwinnett Research institute, LLC, Buford, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Gwinnett Biomedical Research, Lawrenceville, Georgia
  - DC Research Work, Marietta, Georgia
  - Southeast Lung Associates Research, Rincon, Georgia
  - Saltzer Medical Group, Nampa, Idaho
  - PMG Research of Christie Clinic, Champaign, Illinois
  - Medical and Procedural Specialists of Illinois, LLC, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Community Hospital of Anderson and Madison County, Inc., Anderson, Indiana
  - Heartland Research Associates, LLC-An AMR Company, Augusta, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - MedStar Shah Medical Group, Hollywood, Maryland
  - Lahey Clinic, Inc, Burlington, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Somnos Laboratories, Lincoln, Nebraska
  - Creighton University, Omaha, Nebraska
  - Virtua Health, Inc, Marlton, New Jersey
  - Pulmonary Ultimate Research Experience, LLC (PURE, LLC), Toms River, New Jersey
  - Albany Medical College MC-91, Albany, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Northwell Health, New Hyde Park, New York
  - American Health Research, LLC, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Gastonia Pharmaceutical Research, Gastonia, North Carolina
  - Pulmonix, LLC, Greensboro, North Carolina
  - Hickory Research Center DBA Research Carolina of Hickory, Hickory, North Carolina
  - Coastal Carolina Health Care, New Bern, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Clinical Trial Developers, Inc., Milford, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - The Oregon Clinic, PC, Portland, Oregon
  - Chest Diseases of Northwestern PA, Erie, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Anderson Pharmaceutical Research, LLC, Anderson, South Carolina
  - Charletson Research Institute, Charleston, South Carolina
  - The Medical University of South Carolina, Charleston, South Carolina
  - VitaLink Research--Gaffney (Gaffney Pharmaceutical Research, LLC), Gaffney, South Carolina
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - Clinical Research of Rock HIll, Rock Hill, South Carolina
  - VitaLink Research-Rock Hill, Rock Hill, South Carolina
  - South Carolina Pharmaceutical Research, LLC, Spartanburg, South Carolina
  - Union Pharmaceutical Research, Union, South Carolina
  - Houston Pulmonary Sleep and Allergy Associates, Cypress, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Envision Cancer Care, LLC, Laredo, Texas
  - Renovatio Clinical Consultants, LLC, The Woodlands, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - William S. Middleton Memorial Veterans Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol, informed consent form, and clinical study report will also be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requesors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.